CLINICAL TRIAL: NCT02854917
Title: Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: A Randomized Controlled Trial: Further Study, Health Outcome
Brief Title: Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: Health Outcome
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Forest Laboratories (Industry); Fisher Center for Alzheimer's Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 12444
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Memantine Alone: 10 subjects who previously participated in the "Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: A Randomized Controlled Trial" study will be enrolled in this cohort. These subjects received memantine for a period of 28 weeks.
- Memantine plus Individualized Management of AD: 10 subjects who previously participated in the "Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: A Randomized Controlled Trial" study will be enrolled in this cohort. These subjects received memantine plus individualized management of AD for a period of 28 weeks.

SUMMARY:
This study is a retrospective review of the data collected in a previously completed randomized, controlled trial (RCT) entitled "Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: A Randomized Controlled Trial" (NCT00120874). As part of the previously completed RCT, participants with Alzheimer's Disease (AD) were randomly placed into one of two groups: memantine, or memantine plus an individualized management program consisting of home visits, educational sessions for caregivers, and a caregiver support group. Participants received the study intervention for 28 weeks; study follow-up lasted for 52 weeks.

The collected data from the existing study books from the 28 week treatment portion of the RCT will be carefully examined with respect to each of the research questions for the present retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in the "Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: A Randomized Controlled Trial" study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will only include data from previous participants in the "Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: A Randomized Controlled Trial" study. In total, 20 participants completed the previous RCT and will have their data included in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Total number of prescription medications taken throughout the study | 28 weeks
Total number of hospitalizations | 28 weeks
The total number of new medical conditions | 28 weeks
Total number of days of hospice care | 28 weeks

SECONDARY OUTCOMES:
Total number of psychotropic medications used | 28 weeks
Total number of increases in psychotropic medications | 28 weeks
Total number of decreases in psychotropic medications | 28 weeks
Total number of cardiac medications taken during the study | 28 weeks
Total number arthritic and anti-inflammatory medications taken during the study | 28 weeks
Total number of analgesic medications taken during the study | 28 weeks
Total number of days hospitalized during the study | 28 weeks
Reasons for hospitalizations and hospital diagnoses during the study | 28 weeks
  This endpoint will be examined qualitatively; no statistical analysis will be performed but the data will be compiled and reported for illustrative purposes
Total number of tests and procedures performed during the hospitalizations | 28 weeks
Changes in Functional Assessment Staging Disability Score (FAST-DS) at subsequent study visits post hospitalization | 28 weeks
  The FAST-DS assesses the magnitude of progressive functional deterioration by identifying characteristic progressive disabilities in participants with AD. Scores range from 1.0 (normal) to 7f (severe loss of ability, not even able to hold up head independently). Scores are made up of stages (1 through 7) and substages (from a to e for stage 6; from a to f for stage 7). The following scoring for substages is applied: 6a=6.0, 6b=6.2, 6c=6.4, 6d=6.6, 6e=6.8, 7a=7.0, 7b=7.2, 7c=7.4, 7d=7.6, 7e=7.8, 7f=8.0. Additionally, non-consecutive deficits are noted and scored as follows: full stage non-consecutive deficit=1.0, non-consecutive substage deficit=0.2.
  The overall FAST-DS score = (FAST Stage Score) + (Each Non-Consecutive FAST disability scored as described)
Time to death | 28 weeks
Cause of death | 28 weeks
  This endpoint will be examined qualitatively; no statistical analysis will be performed but the data will be compiled and reported for illustrative purposes
Caregiver training and support in relation to mortality | 28 weeks
  This endpoint will be examined qualitatively; no statistical analysis will be performed but the data will be compiled and reported for illustrative purposes
Differences in rate of fecal incontinence | 28 weeks
Differences in rate of urinary incontinence | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry Reisberg, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ClinicalTrials.gov record for the previously completed RCT — https://clinicaltrials.gov/show/NCT00120874